CLINICAL TRIAL: NCT05337956
Title: Evaluation of the Ultrasound-guided Erector Spinae Plane Block Using Catheter for Postoperative Analgesia in Video-assisted Thoracoscopy: A Prospective, Randomized, Controlled Clinical Trial
Brief Title: Ultrasound-guided Erector Spinae Plane Block Using Catheter for Video-assisted Thoracoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Security Forces Hospital (Other)
Responsible Party: Principal Investigator, Anwar ul Huda, Consultant Anesthesia, Security Forces Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SFH-ESPB
Record Dates: First submitted 2022-03-12; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Post Operative Pain; Opioid Use
Keywords: erector spinae block; Video-assisted thoracoscopy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ESPB catheter group (Active Comparator): Patient in this group will receive ESP block
  Interventions: Procedure: Erector spinae plane block catheter
- Control group (No Intervention): Patient in this group will not receive any block

INTERVENTIONS:
Procedure: Erector spinae plane block catheter — All ESP blocks will be performed in lateral position after general anesthesia induction. ESPB will be performed under ultrasonographic guidance using a linear 6- to 10-MHz ultrasound probe. The linear ultrasound transducer will be placed in a longitudinal parasagittal orientation 3 cm lateral to the T6-10 spinous process. The erector spinae muscles will be identiﬁed superﬁcial to the tip of the transverse process. A 21-gauge 10-cm needle will be inserted using an in-plane superior-to-inferior approach or an out of plane approach. The tip of the needle will be placed into the fascial plane on the deep (anterior) aspect of erector spinae muscle. The location of the needle tip will be conﬁrmed by visible ﬂuid spread lifting erector spinae muscle oﬀ the bony shadow of the transverse process on Ultrasonographic imaging. A total of 10-15 ml of 0.2% ropivacaine will be injected each side. A catheter will then be placed leaving 5 cm in place.
  Arms: ESPB catheter group

SUMMARY:
Different modalities ranging from patient controlled analgesia (PCA) to different regional blocks have been used to control postoperative pain after thoracic surgeries. Thoracic epidural analgesia and paravertebral blocks are effective modes of pain relief but have the risks of severe complications and side effects which include severe hypotension, nerve injury or spinal cord injury, vascular injury and pleural injury etc.

Erector spinae plane block (ESPB) is relatively new regional technique which was described by Forero et al in 2016. Several studies have demonstrated an effective role of ESPB in controlling pain for thoraco-abdominal surgeries which include breast surgery, thoracic surgery and upper GI laparoscopy. Shim et al in their study showed that ESPB significantly reduced pain score in first 6 hours postoperatively in patients who underwent VATS. The aim of this study is to evaluate the eﬀect of ESPB using catheter on postoperative 24 hours opioid consumption in video-assisted thoracoscopy (VATS)

DETAILED DESCRIPTION:
Video-assisted thoracoscopic surgery (VATS) is more commonly used technique nowadays in thoracic surgery. This technique is associated with lesser postoperative pain, better postoperative pulmonary function, decreased mortality and shorter hospital stay. However, patients can have severe and prolonged postoperative pain following VATS. Homma et al reported that 18.8 % of patients have persistent pain following VATS. Acute postoperative pain is considered to be one of strong predictor of persistent pain postoperatively.

Different modalities ranging from patient controlled analgesia (PCA) to different regional blocks have been used to control postoperative pain after thoracic surgeries. Thoracic epidural analgesia and paravertebral blocks are effective modes of pain relief but have the risks of severe complications and side effects which include severe hypotension, nerve injury or spinal cord injury, vascular injury and pleural injury etc.

Erector spinae plane block (ESPB) is relatively new regional technique which was described by Forero et al in 2016. Several studies have demonstrated an effective role of ESPB in controlling pain for thoraco-abdominal surgeries which include breast surgery, thoracic surgery and upper GI laparoscopy. Shim et al in their study showed that ESPB significantly reduced pain score in first 6 hours postoperatively in patients who underwent VATS. The objective of this study is to investigate the role of ESPB using catheter in reducing opioid requirements in first 24 hours after VATS.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18-70 years, ASA 1 to 3 undergoing video-assisted thoracoscopy

Exclusion Criteria:

* Patient refusal, Contraindication to regional anesthesia, Allergy to local anesthesia, bleeding diathesis, use of anticoagulants or corticosteroids, inability to operate PCA, psychiatric disorders or use of psychiatric medications, conversion to open thoracotomy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
24 hours opioid consumption | 24 hours
  How much opioid (morphine equivalents) in milligrams was consumed in 24 hours after surgery

SECONDARY OUTCOMES:
Numerical rating score (NRS) pain score at 15 minutes, 30 minutes, 1 hour, 2 hours, 6 hours, 12 hours, 18 hours and 24 hours after surgery both at rest and when coughing | first 24 hours
  Pain score measure by NRS pain score in postoperative period
Postoperative nausea and vomiting | 24 hours
  The incidence and severity of postoperative nausea and vomiting
Postoperative shoulder pain | 24 hours
  Any complaint of Pain in shoulder in postoperative period will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Security Forces Hospital Program, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
It will be provided on request
Supporting Information: Study Protocol
Time Frame: 2 months
Access Criteria: On request